CLINICAL TRIAL: NCT04415762
Title: A Multicenter Italian and Spanish Observational Registry on Patients Affected by Spontaneous Coronary Artery Dissection (SCAD)
Brief Title: Spontaneous Coronary Artery Dissection Registry (DIssezioni Spontanee COronariche ITalian-SPAnish)
Acronym: DISCO-IT/SPA
Status: Completed | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, Principal Investigator, San Luigi Gonzaga Hospital
Other Study IDs: 001-2020
Record Dates: First submitted 2020-05-20; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Spontaneous Coronary Artery Dissection
Keywords: Spontaneous coronary artery dissection; SCAD
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will investigate the clinical features, acute management and follow up of patients affected by spontaneous coronary artery dissection

DETAILED DESCRIPTION:
Spontaneous Coronary Artery Dissection is now being increasingly studied as it is getting more and more relevant as a cause of ACS. Its management is currently a matter of debate due to the absence of RCT and even the trigger events related to this kind of infarction are still unclear. Notably, the benefits from the use of the antiplatelet medications that prolong bleeding time for a condition whose primary pathophysiology may be an intramural bleed are under discussion.

Hence, the targets pursued by our study may be essentially distinguished in five main points:

1. To assess the characteristics of SCAD patients highlighting the predisposing and precipitating factors related to the acute event
2. To analyze clinical presentation and management of spontaneous coronary dissections in terms of therapeutic approach in the acute phase (conservative therapy vs revascularization)
3. To evaluate the incidence of SCAD recurrence and of major adverse cardiovascular events (MACEs) at follow-up
4. To analyze the impact of a single antiplatelet therapy (SAPT) over the dual one (DAPT) along with the impact of different P2Y12i regimens on acute and long-term prognosis
5. To evaluate impact of different angiographic SCAD type on outcome

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a novel diagnosis of Spontaneous Coronary Artery Dissection (SCAD)

Exclusion Criteria:

* Age <18 year old or inability to provide Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a novel diagnosis of Spontaneous Coronary Artery Dissection (SCAD) confirmed by core-lab analysis of coronary angiograms and other intravascular imaging available
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Major Cardiovascular Cardiac Events (a composite of all-cause of death, non-fatal Myocardial Infarction (MI) and any unplanned revascularization either percutaneous or surgical) | 12 months
  Major Cardiovascular Cardiac Events occurring within 12 months

SECONDARY OUTCOMES:
all-cause of death | 12 months
  all-cause of death
non-fatal Myocardial Infarction (MI) | 12 months
  non-fatal Myocardial Infarction (MI)
any unplanned revascularization either percutaneous or surgical | 12 months
  any unplanned revascularization either percutaneous or surgical

OTHER OUTCOMES:
Major Cardiovascular Cardiac Events (a composite of all-cause of death, non-fatal Myocardial Infarction (MI) and any unplanned revascularization either percutaneous or surgical) in Single vs Double Antiplatelets therapies in conservatively treated SCAD | 12 months
Major Cardiovascular Cardiac Events (a composite of all-cause of death, non-fatal Myocardial Infarction (MI) and any unplanned revascularization either percutaneous or surgical) in Medical treatment vs PCI treated SCAD | 12 months
Major Cardiovascular Cardiac Events (a composite of all-cause of death, non-fatal Myocardial Infarction (MI) and any unplanned revascularization either percutaneous or surgical) in different angiographics SCAD type. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Cerrato, MD, Principal Investigator — San Luigi Gonzaga University Hospital, Orbassano,Turin, Italy

REFERENCES:
- [Derived] Benenati S, Giacobbe F, Zingarelli A, Macaya F, Biole C, Rossi A, Pavani M, Quadri G, Barbero U, Erriquez A, Aranzulla T, Cavallino C, Buccheri D, Rolfo C, Patti G, Gonzalo N, Chinaglia A, Musumeci G, Escaned J, Varbella F, Cerrato E, Porto I; DISCO Collaborators. Interventional Versus Conservative Strategy in Patients With Spontaneous Coronary Artery Dissections: Insights From DISCO Registry. Circ Cardiovasc Interv. 2023 Jun;16(6):e012780. doi: 10.1161/CIRCINTERVENTIONS.122.012780. Epub 2023 Jun 1. PMID 37259861
- [Derived] Cerrato E, Giacobbe F, Quadri G, Macaya F, Bianco M, Mori R, Biole CA, Boi A, Bettari L, Rolfo C, Ferrari F, Annibali G, Scappaticci M, Pavani M, Barbero U, Buccheri D, Cavallino C, Lombardi P, Bernelli C, D'Ascenzo F, Infantino V, Gambino A, Cinconze S, Rognoni A, Montagna L, Porto I, Musumeci G, Escaned J, Varbella F; DISCO Collaborators. Antiplatelet therapy in patients with conservatively managed spontaneous coronary artery dissection from the multicentre DISCO registry. Eur Heart J. 2021 Aug 31;42(33):3161-3171. doi: 10.1093/eurheartj/ehab372. PMID 34338759